CLINICAL TRIAL: NCT05544292
Title: Rheumatic IMmune-Related Adverse Events in Patients Treated With Immune Check Point Inhibitors - a Prospective Observational Study
Brief Title: Rheumatic IMmune-Related Adverse Events in Patients Treated With Immune Check Point Inhibitors
Acronym: RIMRA
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other); Alesund Hospital (Other); University Hospital of North Norway (Other); Hospital of Southern Norway Trust (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: DS 00469
Record Dates: First submitted 2022-08-17; First posted 2022-09-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Immune-related Adverse Event
Keywords: arthritis; check point inhibitor; irAE
MeSH Terms: conditions — Arthritis | interventions — Anti-Inflammatory Agents; Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and whole blood samples are collected at baseline and after 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antiinflammatory/DMARDs — Antiinflammatory/DMARDs

SUMMARY:
RIMRA is a prospective, longitudinal, observational study including patients with de novo symptoms of rheumatic disease or a flare of established rheumatic disease after treatment with an immune check point inhibitor. The aim of the study is to describe the clinical presentation, disease course and outcome of rheumatic irAEs in patients treated with immune check point inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* De novo symptoms of rheumatic disease or a flare of established rheumatic disease after >/= 1 dose of treatment with an immune check point inhibitor
* Adult patients (> 18 years)
* Subject capable of understanding and signing an informed consent form

Exclusion Criteria:

• Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred with symptoms of a rheumatic condition after cancer treatment with a check point inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Swollen joint count | 1 year follow-up
  Numbers (0-66)

SECONDARY OUTCOMES:
C reactive protein | 1 year
  mg/L
Proportion of pateints with arthritis after one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marte S Heiberg, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (5):
- Norway (5):
  - Ålesund Hospital, Ålesund
  - Hospital of Southern Norway Trust, Kristiansand
  - Levanger Hospital, Levanger
  - Diakonhjemmet Hospital, Oslo
  - University Hospital of North Norway, Tromsø